CLINICAL TRIAL: NCT00869271
Title: Postoperative folfox4 Only vs folfox4 Plus TAC in the Treatment Unresectable Liver Metastasis of Colorectal Cancer: a Randomized,Prospective,Control Trial
Brief Title: Postoperative Folfox4 Only Versus Folfox4 Plus Transhepatic Arterial Chemotherapy (TAC) in the Treatment Unresectable Liver Metastasis of Colorectal Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Xujianmin, Zhongshan hospital, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-01
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Unresectable Liver Metastasis of Colorectal Cancer
Keywords: liver metastasis; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Triamcinolone; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): folfox4 chemotherapy was done within 28 days after primary surgery. Per 3 weeks, patients will receive one cycle. After 3 cycles, patients will received transhepatic arterial chemotherapy(TAC) using oxaliplatin, fudr and mmc. Then begin folfox4 again.
  Interventions: Procedure: tac + folfox4
- 2 (Active Comparator): folfox4 chemotherapy was done within 28 days after primary surgery. Per 3 weeks, patients will receive one cycle.
  Interventions: Procedure: Folfox4

INTERVENTIONS:
Procedure: tac + folfox4 — tac: oxaliplatin 100mg + fudr 1g + mmc 10mg
  folfox4
  Folfox4 chemotherapy was done within 28 days after primary surgery. Per 3 weeks, patients will receive one cycle. After 3 cycles, patients will received transhepatic arterial chemotherapy(TAC) using oxaliplatin, fudr and mmc. Then begin folfox4 again.
  Arms: 1
Procedure: Folfox4 — folfox4
  Folfox4 chemotherapy was done within 28 days after primary surgery. Per 3 weeks, patients will receive one cycle
  Arms: 2

SUMMARY:
The purpose of this study is to investigate whether TAC plus FOLFOX4 are able to improve resection rate and overall survival in patients receiving primary colorectal tumor resection than given FOLFOX4 only.

DETAILED DESCRIPTION:
We administered three cycles FOLFOX4 plus on TAC (oxaliplatin, FUDR and MMC) or FOLFOX4 only to primary colorectal tumor resected patients with unresected liver metastasis. The study endpoints were resection rate of liver metastasis, progression-free survival, overall survival as evaluated by intent-to-treat analysis.

ELIGIBILITY:
Inclusion Criteria:

* age < 75 years with histologically proven adenocarcinoma of the colon or rectum
* no severe major organ dysfunction
* WHO performance status of 0 or 1
* no prior cancer therapy
* with measurable unresectableliver metastasis
* without other metastasis

Exclusion Criteria:

* age >= 75
* severe major organ dysfunction
* WHO performance status of >1
* prior cancer therapy
* with other metastasis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2005-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
overall survival | 5 years after diagnosis

SECONDARY OUTCOMES:
progression free survival | 5 years after diagonsis

CONTACTS AND LOCATIONS:
Overall Officials: jianmin xu, MD, PHD, Study Director — department of general surgery, zhongshan hospital, fudan university
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China